CLINICAL TRIAL: NCT05055726
Title: Phase IV Study on the Feasibility of a Preventative/Therapeutic Approach With Benzydamine Oromucosal Solution in Radiation-induced Oral Mucositis (OM) in Patients With Head and Neck Cancer (HNC)
Brief Title: Benzydamine Oromucosal Solution in Oral Mucositis (BOOM)
Acronym: BOOM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030(Z)WO19247; 2020-003306-32 (EudraCT Number)
Record Dates: First submitted 2021-06-23; First posted 2021-09-24 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Radiation-Induced Mucositis; Head and Neck Cancer
Keywords: oral mucositis; radiation therapy; head and neck cancer; mouthwash; oromucosal solution; benzydamine
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis | interventions — Benzydamine

STUDY DESIGN:
Intervention Model Description: multicenter, international, open label, single-group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benzydamine Hydrochloride 0.15% w/v oromucosal solution (Experimental): Benzydamine Hydrochloride 0.15% w/v oromucosal solution (mouthwash), Angelini Pharma S.p.A., is assigned to the patients for radiation-induced oromucositis.
  The patients take at home 15 ml (1 tablespoon) of concentrated or diluted (with water) mouthwash 2-3 times a day, but not more than 5 times a day, washing the mouth and throat for 20-30 seconds, according to the Investigator's indications and the local product's SmPC.
  In Hungary, the therapy should started with diluted product (15 ml of water + 15 ml of concentrated solution). After that, gargling can be continued with 15 ml (1 tablespoon) of concentrated mouthwash, generally 2-3 times a day, but not more than 5 times a day.
  In Poland, the solution is used 2 to 3 times daily; at a single time, it should be used approximately 15 ml of concentrated or diluted mouthwash with a small amount of water and wash the mouth and throat for 20 to 30 seconds.
  Interventions: Drug: Benzydamine Hydrochloride 0.15% w/v oromucosal solution

INTERVENTIONS:
Drug: Benzydamine Hydrochloride 0.15% w/v oromucosal solution — Benzydamine Hydrochloride 0.15% w/v oromucosal solution (mouthwash), Angelini Pharma S.p.A.

SUMMARY:
The aim of the present study is to collect data on the feasibility of a preventative/therapeutic approach of radiation-induced oral mucositis with benzydamine oromucosal solution (mouthwash) in patients with head and neck cancer.

DETAILED DESCRIPTION:
This is a phase IV clinical study whose aim is to collect data on the feasibility of a preventative/therapeutic approach of radiation-induced oral mucositis with benzydamine oromucosal solution (mouthwash) in patients with Head and Neck cancer.

Benzydamine mouthwash is considered the gold standard among anti-inflammatory agents in the management of oral mucositis in cancer patients.

The 2014 mucositis guidelines recommended benzydamine mouthwash for the prevention of radiation-induced oral mucositis among Head and Neck Cancer patients treated with moderate doses of radiation therapy. The updated 2019 guidelines not only confirm the existing guidelines proving new evidences, but also recommend to use benzydamine as preventative treatment of radiation-induced Oromucositi among Head and Neck Cancer. patients treated with radiation therapy with/without systemic concurrent treatments and confirm benzydamine mouthwash as the only anti-inflammatory agent with evidence in prevention of oral mucositis to date.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any ethnic origin ≥18 years of age.
* Patients diagnosed with stage III or IV Head and Neck cancer (histologic or cytologic diagnosis), according to VIII AJCC staging system, who are candidate and are about to start RT, with or without concomitant CT, with curative intent, either with exclusive or postoperative intent.
* Eastern Cooperative Oncology Group (ECOG) performance status with a score of 0, or 1, or 2.
* Patients legally capable of giving their consent to participate in the study and available to sign and date the written informed consent and the Declaration of consent for the processing of personal data.
* Women of childbearing potential or with no menses for a period < 12 months must have a negative pregnancy test at Visit 0 and have to agree not to start a pregnancy from the signature of the informed consent up to the end of the study, using an appropriate birth control method, such as combined oestrogen-progestin containing hormonal contraceptives (e.g., oral, injectable, transdermal), progestin-only hormonal contraceptives (e.g., oral, injectable, implantable), intrauterine device (IUD) or Intrauterine hormone-releasing System (IUS) in combination with male condom, bilateral tubal occlusion, vasectomised partner, sexual abstinence. The following definitions will be considered:

  * Woman of childbearing potential (WOCBP): i.e., fertile, following menarche and until becoming post-menopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Exclusion Criteria:

* Patients with reported allergy to benzydamine or another component of the formulation used.
* Any contraindications listed in the local product's Summary of Product Characteristics (SmPCs).
* Patients with prior head and neck RT (in the previous 6 months), or patient who received a palliative treatment.
* Patients with distant metastatic disease and/or severe cognitive impairment and/or clinically symptomatic brain metastases and/or patients with significant comorbid conditions.
* Patients with mucositis due to other medical conditions (e.g., gastro-oesophageal reflux, autoimmune disease, etc.).
* Patients who use other oromucosal products (over the counter or prescription) for the same disease.
* Prescription of other rinses (anaesthetics like "magic mouthwashes" or others), except from sodium bicarbonate rinses.
* Use of chlorhexidine, other anti-inflammatory mouthwashes solutions, misoprostol, granulocyte macrophage colony-stimulating factor (GM-CSF) and sucralfate gel.
* Employment of antifungal or antibiotic drugs as prophylaxis for mucositis; any therapeutic use in case of overt clinical infections is allowed.
* Patients treated with other therapies that can cause mucositis, except for the therapies for their primary condition.
* Patients treated with any topical anti-inflammatory/analgesic products for the mucositis.
* Any other product that can interfere with the evaluation of pain or inflammatory state, according to the Investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Number of responders | Up to 7 weeks
  The effectiveness of benzydamine oromucosal solution (mouthwash) in the prevention/tratment of radiation-induced oral mucositis in Head and Neck cancer patients is evaluated as the number of responders, expressed in percentage, defined as the number of head and neck cancer patients with oral mucositis pain intensity <5 in the Numeric Rating Scale.

SECONDARY OUTCOMES:
Number of compliant patients to Benzydamine treatment. | Up to 7 weeks
  The compliance to the treatment is calculated at the end of the study. A patient is considered compliant to the benzydamine treatment if he/she takes ≥80% of the total dose assigned by the Investigator.
Change score in the World Health Organization oral mucositis grading scale. | Up to 7 weeks
  The severity of oral mucositis is evaluated using the World Health Organization (WHO) oral mucositis grading scale.
  The Investigator gives a score corresponding to the grade of mucositis of the patient, from "0" = "None" to "4" = "Life-threatening", "Oral alimentation impossible".
Number of days of duration of severe oral mucositis. | Up to 7 weeks
  The duration of severe oral mucositis (grade 3 or 4 on the World Health Organization oral mucositis grading scale) is assessed.
Time of onset of severe oral mucositis. | Up to 7 weeks
  Time of onset of severe oral mucositis (grade 3 or 4 on the World Health Organization oral mucositis grading scale) is assessed.
Percentage change in body weight | Up to 7 weeks
  The percentage change in body weight from baseline is assessed.
Number of days of duration of Radiotherapy/Chemotherapy | Up to 7 weeks
  Radiotherapy/Chemotherapy is assessed as number of days of duration of therapy.
Number of days of discontinuation of Radiotherapy/Chemotherapy | Up to 7 weeks
  Radiotherapy/Chemotherapy is assessed in terms of days of therapy discontinuation.
Dose modifications of Radiotherapy/Chemotherapy | Up to 7 weeks
  Radiotherapy/Chemotherapy is evaluated as dose modifications of therapy.
Delays in Radiotherapy/Chemotherapy | Up to 7 weeks
  Radiotherapy/Chemotherapy is evaluated as days of delay in therapy.
Number of days of hospitalization. | Up to 7 weeks
  The healthcare resources consumed in terms of number of days of hospitalization due to oral mucositis are evaluated.
Change in QoL (EORTC QLQ C-30) from baseline | Up to 7 weeks
  The health-related quality of life is measured using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C-30)
Change in QoL (EORTC QLQ-H&N35) from baseline | Up to 7 weeks
  The health-related quality of life is measured using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck (EORTC QLQ-H&N35).
Number and type of opioid analgesics | Up to 7 weeks
  The use of opioid analgesics prescribed for oral mucositis pain is assessed.
Frequency of adverse events | Up to 7 weeks
  AEs occurred during a clinical trial are assessed by the Investigator in terms of seriousness and relationship with the investigational product.

CONTACTS AND LOCATIONS:
Locations (10):
- Hungary (6):
  - Orszagos Onkologiai Intezet, Gyogyszertar, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Intezeti Gyogyszertar, Debrecen
  - Petz Aladar Egyetemi Oktato Korhaz, Intezeti Gyogyszertar,, Győr
  - Somogy Megyei Kaposi Mor Oktato Korhaz - Eszaki Tomb, 1. Emelet, 4. Szarny, Klinikai - Vizsgalati Egyseg., Kaposvár
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Josa Andras Oktatokorhaz Klinikai Kutatasi Osztaly, Nyíregyháza
  - Csolnoky Ferenc Korhaz, Onkologiai Centrum Sugarterapias Osztaly, Veszprém
- Poland (4):
  - Centrum Onkologii im. Prof. Franciszka Łukaszczyka Apteka Szpitalna, Bydgoszcz
  - Szpitale Pomorskie Sp. z o. o.,, Gdynia
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii I Traumatologii im. M. Kopernika w Lodzi, - Lódzkie, Lodz
  - Mazowiecki Szpital Wojewódzki im. św. Jana Pawła II w Siedlcach -, Siedlce